CLINICAL TRIAL: NCT02892773
Title: A Randomized Controlled Trial Comparing the Effectiveness of Lung Expansion Therapy Following Upper Abdominal Surgery in Adult Human Subjects
Brief Title: Comparing the Effectiveness of Lung Expansion Therapy in Adult Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Draeger Medical, Inc (Industry)
Responsible Party: Principal Investigator, Daniel D Rowley, MSc RRT-ACCS, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19029
Record Dates: First submitted 2016-08-28; First posted 2016-09-08 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Atelectasis
Keywords: electrical impedance tomography; incentive spirometry; EzPAP; lung volume; atelectasis; positive airway pressure; pulmonary complication; abdominal surgery; end-expiratory lung volume
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant and Care Provider will be masked from electrical impedance tomography distribution of ventilation recording during lung expansion therapy to reduce risk of performance bias.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incentive Spirometry Group (Other): * Participant will be asked to take 10 deep breaths through the mouthpiece of an incentive spirometer, followed by a 60 second pause.
  * This cycle will be repeated two more times.
  * A Respiratory Therapist will coach participants three times per day.
  * Each duration of Incentive Spirometry will last about 15 minutes.
  Interventions: Device: Incentive Spirometry
- EzPAP® Positive Airway Pressure Group (Active Comparator): * Participant will be coached by a Respiratory Therapist to breathe through the mouthpiece of an EzPAP® device for 10 breaths, followed by a 60 second pause.
  * This cycle will be repeated two more times.
  * The Respiratory Therapist will coach participants three times per day.
  * Each duration of EzPAP® therapy will last about 15 minutes.
  Interventions: Device: EzPAP® Positive Airway Pressure

INTERVENTIONS:
Device: Incentive Spirometry — A respiratory therapist will provide instruction on Incentive Spirometry (I.S.) procedure performance before supervised therapy and monitoring begins.
  * Study participants will be asked to take 10 deep breaths through the I.S.'s mouthpiece, followed by a 60 second pause.
  * The 10-breath cycle will be repeated 3 times per therapy session.
  * Each I.S. therapy session will last about 15 minutes, 3 times per day.
  * Lung monitoring and deep breathing measurements will occur during a scheduled I.S. sessions on day 1, 3, and 5 after surgery.
  Arms: Incentive Spirometry Group
Device: EzPAP® Positive Airway Pressure — A respiratory therapist will provide instruction on EzPAP® procedure performance before supervised therapy and monitoring begins.
  * Study participants will be asked to breathe normally through the EzPAP® device's mouthpiece for 10 breaths, followed by a 60 second pause.
  * The 10-breath cycle will be repeated 3 times.
  * Each EzPAP® therapy sessions will last about 15 minutes, 3 times per day.
  * Lung monitoring will occur during a scheduled EzPAP® sessions on day 1, 3, and 5 after surgery.
  Arms: EzPAP® Positive Airway Pressure Group

SUMMARY:
The purpose of this study is to better understand how air is spread throughout study participants' lungs after abdominal surgery by comparing two lung inflation treatments:

1. Incentive Spirometry (I.S.) lung expansion therapy
2. EzPAP® lung expansion therapy.

Lung expansion therapy is routinely used after upper abdominal surgery. Taking deep breaths after surgery helps lungs to stay inflated. At the University of Virginia, it is at the physician's discretion as to which treatment will be used to help with deep breathing lung inflation therapy after surgery. The investigators would like to know which of the lung inflation therapies is better at helping inflate participants' lungs.

The investigators will be using a device called Electrical Impedance Tomography (EIT) to measure how effectively air spreads in participants' lungs. This device is not currently approved by the Food and Drug Administration (FDA) for the purpose used in this study, and therefore, it is considered investigational.

Investigators are inviting eligible participants to consider participating in this study because doctors order Incentive Spirometry as a standard of care following upper abdominal surgery. Information gained from monitoring how air is spread throughout participants' lungs will help investigators to determine if there is a clinical difference and benefit when comparing Incentive Spirometry and EzPAP lung expansion therapies.

DETAILED DESCRIPTION:
Investigators will use a convenience sampling scheme to identify potential study participants. Documentation of informed consent will be recorded. Electrical Impedance Tomography (EIT), which provides non-invasive and radiation free monitoring, will be used to monitor and measure regional distribution of ventilation during Incentive Spirometry (I.S.) and EzPAP® lung expansion therapy. The PulmoVista 500 EIT device has a reported high patient safety profile and poses minimal patient risk.

The potential benefit for study participants will not be realized directly since the investigators' aim is to only monitor regional distribution of ventilation in response to I.S. or EzPAP® lung expansion therapy. While I.S. is considered to be a standard of post-operative care, there is low quality evidence documenting I.S. effectiveness in preventing pulmonary complications after upper abdominal surgery.

Loss of dorsal lung volume (i.e., atelectasis) is an example of a post-operative pulmonary complication. EzPAP® is a lung expansion therapy that is used as an alternative to I.S. lung expansion therapy for increasing dorsal regional lung volume (i.e., Functional Residual Volume [FRC]) in an effort to prevent or reverse atelectasis. When expiratory positive airway pressures of 5, 10, and 15 cmH2O was administered to a small group of healthy human subjects, medical researchers identified that a positive pressure of 15 cmH2O was associated with the greatest FRC increase when compared to zero pressure and baseline FRC measurements.

While study participants may not benefit directly from this study, investigators anticipate that important information will be gained from EIT monitoring of regional distribution of ventilation. Future upper abdominal post-operative surgical patients may benefit from this study's findings as investigators hope to advance clinical understanding associated with these therapies with use of EIT.

Procedure set-up and device calibration will occur according to Draeger provided PulmoVista 500 EIT training and operation manual instructions:

* Study participant preparation

  * Investigators will assess the participant's thorax to ensure that the skin's surface is free of body fluids that may prevent or impede electrode contact. Skin surface will be wiped clean with a dry cloth if necessary.
  * Investigators will select an electrode belt and respective patient cable sizes after measuring participant's chest circumference with paper measurement tape placed across the midclavicular line at intercostal space 4 -5. Electrode belt size will be selected according to chest circumference measurement.
  * A patient cable of the same electrode belt size will be selected and connected to the electrode belt before connection to participant. Investigators will align and snap connect the patient cable snaps over the electrode belt studs by aligning respective snaps and studs in ascending numerical order from 1 to 16 .
  * A light spray of water may be applied to the black electrode surface on the electrode belt before it is applied to participant if natural moisture from the skin does not result in sufficient conductivity between the skin and electrodes.
* Investigators will attach an electrode belt and reference electrode to participant while they are lying supine in bed. Participant's head of bed will be positioned at 45-degrees.

  * The electrode belt/cable combination will be attached around the thorax of each participant at the level of the 4th - 5th intercostal space, unless mammary tissue prevents this site of application. An alternative application site will be located immediately below the mammary tissue if necessary. Left to right belt orientation will be maintained with color coded patient cable ports signifying left and right side.
  * Investigators will snap the electrode belt closed after verifying proper belt position. The belt's black electrodes should have close contact with the study participant's skin at this point.
  * An adhesive ECG electrode will be place on the study participant's right upper abdominal quadrant and then the patient cable reference electrode snap will be attached to the ECG electrode.
  * The patient cable will then be connected to the EIT monitoring device via a color coded trunk cable orientation that aligns with the patient cable left and right orientation
* EIT device calibration and signal check

  * Investigators will initiate a PulmonVista 500 EIT monitoring device calibration each day prior to performing new study participant end-expiratory lung impedance measurements.
  * A skin-electrode signal check will be performed to ensure that a minimum of 15 of 16 electrodes have sufficient contact with the participant's skin surface and signal quality is stable. Investigators will use the following status display and explanation to determine adequacy of electrode contact and signal quality.
* Monitoring sessions and Lung Expansion Therapy procedure

  * Monitoring will be initiated after investigators perform PulmoVista 500 EIT device setup and calibration prior to one of the three scheduled lung expansion therapy sessions on day 1, 3, and 5 (if not discharged from hospital) after surgery.
  * Approximate monitoring/measurement duration is 15-minutes.
* Lung expansion therapies will occur as follows:

  * Participants will be positioned supine in bed or bedside chair with head of bed or bedside chair positioned at 45-degrees.

Incentive Spirometry Procedure Group:

* A respiratory therapist will provide instruction on Incentive Spirometry procedure performance before supervised therapy and monitoring begins.
* Participants will be asked to take 10 deep breaths through the incentive spirometer's mouthpiece, followed by a 60 second pause.
* The 10-breath cycle will be repeated three times with respiratory therapist coaching.
* Each Incentive Spirometry therapy session will last about 15 minutes three times per day.
* EIT monitoring and deep breathing measurements will occur during one of the three scheduled Incentive Spirometry sessions on day 1, 3, and 5 (if not discharged from hospital) after surgery.

EzPAP® Positive Airway Pressure Group:

* A respiratory therapist will provide instruction on EzPAP® procedure performance before supervised therapy and monitoring begins.
* Participants will be asked to breathe normally through the EzPAP® device's mouthpiece for 10 breaths, followed by a 60 second pause.
* The 10-breath cycle will be repeated three times with respiratory therapist coaching.
* Each TID EzPAP® therapy sessions will last about 15 minutes three times per day.
* EIT monitoring and deep breathing measurements will occur during one of the three scheduled Incentive Spirometry sessions on day 1, 3, and 5 (if not discharged from hospital) after surgery.

  • PulmoVista set-up and monitoring sessions will be coordinated in collaboration with each participant's bedside nurse and a respiratory therapist. Initial setup and monitoring commitment time is approximately 15 - 20 minutes.
* Electrical Impedance Tomography lung monitoring and measurements will occur during one of three scheduled EzPAP® therapies on day 1, 3, and 5 (if not discharged from hospital) after surgery. Participants will continue to receive respective lung expansion therapy as ordered three times per day, but without EIT monitoring.

  • Regional distribution of ventilation information will be displayed on the PulmoVista 500 device's main monitoring screen during lung expansion therapy. Clinical staff administering therapy and participants will be blinded from information displayed on the screen's monitor in an effort to reduce performance bias.
* Once lung expansion therapy session has ended, investigators will detach trunk cables from electrode cables, detach reference electrode snap from adhesive ECG electrode, unclamp the electrode belt, and then remove belt from the participant.
* Investigators will inspect the electrode belt contact area to assess for evidence of skin irritation or bruising. Participant's physician will be notified of any significant findings.

  • Displaying changes
* Once the PulmoVista 500 EIT device is removed from participant's room, the investigator will change from main screen view to Display change view. Regional distribution of ventilation information displayed on the PulmoVista 500 EIT device's screen will be used to record pre and post lung expansion therapy end-expiratory lung impedance changes.
* PulmoVista 500 EIT device will be removed participant's room and returned to a storage location outside of patient care areas.

  * Following each EIT to participant interface disconnect, an alcohol, aldehyde, or quaternary ammonium based compound will be soaked on a wipe cloth to disinfect the surfaces of the patient cable, electrode belt, trunk cable, and EIT unit.
  * Participant's head of bed will be returned to original position or to an elevation that is preferred by the participant after therapy and monitoring session is complete.
  * Participant will continue with assigned lung expansion therapy as scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Human subjects 18 - 79 years of age
* Post-operative upper abdominal surgery

Examples:

* Laparotomy
* Biliodigestive anastomosis
* Cholecystectomy
* Enterectomy
* Esophagectomy
* Gastrectomy
* Hepatectomy
* Pancreatectomy
* Unassisted spontaneous breathing

  * Attending surgeon's approval
  * Anticipated post-operative hospital length of stay greater than 3 days
  * Documentation of written informed consent
  * Ability to sign consent

Exclusion Criteria:

* Less than 18 or greater than 79 years of age
* Anticipated post-operative hospital length of stay less than 3 days
* Body mass index > 50
* Excessive chest hair
* Inability to obtain written informed consent
* Inability to follow verbal instructions
* Pregnancy-self reported
* uncontrolled body movements
* Insertion of an artificial airway
* Hemodynamic instability
* Loss of skin integrity at site where EIT electrodes and belt are projected to come into contact (i.e., chest burns, open wounds/lesions, etc…).
* Chest tube or dressings that prohibit placement of EIT electrodes and belt
* Active implants (i.e., cardiac pacemaker, implantable cardioverter-defibrillator [ICD]), diaphragm pacer, or when device compatibility is in doubt.)
* Invasive or non-invasive mechanical ventilation support
* Unstable spinal lesions or fractures
* Untreated pneumothorax
* Active hemoptysis
* Esophageal surgery
* Decision to withhold life-sustaining treatment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-01; Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Ventral and Dorsal end-expiratory lung impedance redistribution of ventilation | Two years
  EIT will be used to measure ventral and dorsal change in end-expiratory lung impedance before and after lung expansion therapy. Ventral and Dorsal lung impedance measurement is displayed on the EIT device as a percent (zero to 100). Investigators will record values into an electronic code book before and after lung expansion therapy. The difference between measured values will be used to quantify ventral and dorsal redistribution of ventilation.
  * Statistical analysis
    * An independent samples t-test or Mann-Whitney U test will be applied to determine if a statistically significant mean difference exists between groups.
    * Data will be reported as mean (SD) and 95% CI or median (IQR) depending upon normality of distribution.
    * Effect size = r (small effect </= 0.1; medium effect = 0.3; Large effect >/= 0.5
    * Alpha set at ≤ 0.05 (two-tailed)

SECONDARY OUTCOMES:
Incidences of post-operative pulmonary complications | Two years
  Investigators will search participant's electronic medical record for documentation of atelectasis, hypoxemia, pneumonia, and acute respiratory failure. Data will be recorded in an electronic code book and total count for respective pulmonary complications will be used to quantify incidence of respective pulmonary complications.
  • Statistical analysis
  * Chi square for independence or Fisher's Exact Probability test will be applied to test for statistical significance.
  * Respective post-operative complication will be reported as frequency (n)
  * Relative Risk and Odds Ratio will be reported for effect size.
  * Alpha set at ≤ 0.05 (two-tailed)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Rowley, MSc RRT-ACCS, Principal Investigator — Pulmonary Diagnostics & Respiratory Therapy Services, University of Virginia Medical Center
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Intend to submit overall study findings to peer reviewed medical journal after study completion.

REFERENCES:
- [Background] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642
- [Background] Fagevik Olsen M, Wennberg E, Johnsson E, Josefson K, Lonroth H, Lundell L. Randomized clinical study of the prevention of pulmonary complications after thoracoabdominal resection by two different breathing techniques. Br J Surg. 2002 Oct;89(10):1228-34. doi: 10.1046/j.1365-2168.2002.02207.x. PMID 12296888
- [Background] Garrard CS, Shah M. The effects of expiratory positive airway pressure on functional residual capacity in normal subjects. Crit Care Med. 1978 Sep-Oct;6(5):320-2. doi: 10.1097/00003246-197809000-00004. PMID 363357
- [Background] Hinz J, Neumann P, Dudykevych T, Andersson LG, Wrigge H, Burchardi H, Hedenstierna G. Regional ventilation by electrical impedance tomography: a comparison with ventilation scintigraphy in pigs. Chest. 2003 Jul;124(1):314-22. doi: 10.1378/chest.124.1.314. PMID 12853539
- [Background] Karsten J, Stueber T, Voigt N, Teschner E, Heinze H. Influence of different electrode belt positions on electrical impedance tomography imaging of regional ventilation: a prospective observational study. Crit Care. 2016 Jan 8;20:3. doi: 10.1186/s13054-015-1161-9. PMID 26743570
- [Background] Lunardi AC, Paisani DM, Silva CCBMD, Cano DP, Tanaka C, Carvalho CRF. Comparison of lung expansion techniques on thoracoabdominal mechanics and incidence of pulmonary complications after upper abdominal surgery: a randomized and controlled trial. Chest. 2015 Oct;148(4):1003-1010. doi: 10.1378/chest.14-2696. PMID 25973670
- [Background] Meier T, Luepschen H, Karsten J, Leibecke T, Grossherr M, Gehring H, Leonhardt S. Assessment of regional lung recruitment and derecruitment during a PEEP trial based on electrical impedance tomography. Intensive Care Med. 2008 Mar;34(3):543-50. doi: 10.1007/s00134-007-0786-9. Epub 2007 Jul 25. PMID 17653529
- [Background] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355
- [Background] Riedel T, Richards T, Schibler A. The value of electrical impedance tomography in assessing the effect of body position and positive airway pressures on regional lung ventilation in spontaneously breathing subjects. Intensive Care Med. 2005 Nov;31(11):1522-8. doi: 10.1007/s00134-005-2734-x. Epub 2005 Sep 30. PMID 16195908
- [Background] Stankiewicz-Rudnicki M, Gaszynski T, Gaszynski W. Assessment of regional ventilation in acute respiratory distress syndrome by electrical impedance tomography. Anaesthesiol Intensive Ther. 2015;47(1):77-81. doi: 10.5603/AIT.2015.0007. PMID 25751294
- [Background] Westerdahl E, Lindmark B, Eriksson T, Friberg O, Hedenstierna G, Tenling A. Deep-breathing exercises reduce atelectasis and improve pulmonary function after coronary artery bypass surgery. Chest. 2005 Nov;128(5):3482-8. doi: 10.1378/chest.128.5.3482. PMID 16304303
- [Derived] Rowley DD, Malinowski TP, Di Peppe JL, Sharkey RM, Gochenour DU, Enfield KB. A Randomized Controlled Trial Comparing Two Lung Expansion Therapies After Upper Abdominal Surgery. Respir Care. 2019 Oct;64(10):1181-1192. doi: 10.4187/respcare.06812. Epub 2019 May 21. PMID 31113857